CLINICAL TRIAL: NCT05356247
Title: Lausanne Trialogue Paradigm - Brief: A Family Systems Model to Address Child Mental Health in a Community Mental Health Setting
Brief Title: Lausanne Trialogue Paradigm - Brief: A Family Model for Child Mental Health in a Community Setting
Acronym: LTP-B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: York University (Other)
Collaborators: University of Lausanne (Other); SickKids Centre for Community Mental Health (SKCCMH) (Unknown)
Responsible Party: Principal Investigator, Heather Prime, Assistant Professor, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-050
Record Dates: First submitted 2022-03-22; First posted 2022-05-02 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Parent-Child Relations; Family Relations; Internet-Based Intervention; Mental Health Issue; Behavioral Problem
Keywords: Child Mental Health; Family Systems; Coparenting; Single arm pre-post design; COVID-19 Family Recovery
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LTP-B Intervention (Experimental): Families will take part in an online semi-structured assessment and video feedback paradigm of family interactions, with an emphasis on co-parenting and parent-child relations.
  Interventions: Behavioral: Lausanne Trialogue Play Brief

INTERVENTIONS:
Behavioral: Lausanne Trialogue Play Brief — The brief treatment program will consist of an LTP family assessment with video feedback to caregivers to address family interaction patterns and child mental health. Families will participate in four sessions conducted online using the Zoom for Healthcare platform. In the first session, families will engage in a family assessment in different groupings that will be recoded on zoom and used later in the treatment. In the second session, taking place one week later, families will take part in a mini assessment to learn more about the difficulties of the child. In the third session, the clinical team will share videos of the family assessment to the parents and discuss the families strengths, concerns, and goals for moving forward. In the fourth session, taking place one month after the third session, families will participate in a check-in session, debriefing the family assessment.
  Other Names: LTP-B

SUMMARY:
The current study is a feasibility pilot of the Lausanne Trialogue Play paradigm Intervention - Brief (LTP-Brief), a family systems therapy implemented in a community mental health setting. We will study the ultrabrief, virtual therapy to assess the feasibility of a future pilot RCT. Feasibility metrics include resource, scientific, and management considerations, as well as an examination of pre-post change in future child and family outcomes of interest.

DETAILED DESCRIPTION:
COVID-19 represents an acute crisis to children's mental health, with potential for long-term consequences. There is evidence for elevated mental health symptomatology in children since the start of the pandemic, with the emergence of stress-related disorders and the exacerbation of pre-existing disorders. Indeed, the pandemic has had detrimental effects on family life due to widespread job loss and financial insecurity, and increases to parental psychological distress, mental illness, and substance use. Social consequences of COVID-19 are expected to have cascading negative effects on child mental health symptoms. Thus, a COVID-19 family recovery program is critically needed, both during and after the pandemic, to manage the current mental health crisis in children and create cascading and sustainable effects for lifelong physical and mental health. The main goal of the the current study is to investigate feasibility of a future pilot and/or main RCT of a brief, virtual mental health treatment program for children and families designed to optimize reach of services. Specifically, the Lausanne Trialogue Play paradigm assessment is a semi-structured assessment of whole family interactions, with emphasis on the co-parenting relationship, which has been used extensively in research settings for assessment and consultative purposes. The current study will assess the feasibility of using the LTP in an assessment-as-treatment model. This brief treatment program, called the LTP-Brief intervention (LTP-B) will consist of a family play assessment (including an LTP assessment) with video feedback to caregivers as a method for promoting change in family interaction patterns. By targeting change across the family system, rather than focusing on specific child mental health symptoms directly, the model addresses upheaval of family life during COVID-19 and has potential to create sustainable improvements in family well-being within a short period of time.

ELIGIBILITY:
Inclusion Criteria:

* The sample will comprise of families referred to the outpatient mental health services at Sick Kids Center for Community Mental Health (SKCCMH), a non-profit children's mental health treatment centre in Toronto, ON, Canada.
* Participants will include children ages 0 months to 15.11 years old, and their caregivers, though the majority will fall in the range of 3- to 14-years-old.
* The first 25 families to be referred to the LTP-B service and who agree to participate in research will be included.

Exclusion Criteria:

* No exclusion criteria beyond what is standard for the clinical service at SKCCMH.

Ages: 0 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
COVID-19-related Family Stressors | Time 0, 3
  Descriptive (no criterion for success): Family Stressor Scale. Minimum score=16, maximum score=48. Higher scores correspond to worse outcomes.
COVID-19-related Family Positive Adaptation | Time 0, 3
  Descriptive (no criterion for success): COVID-19 Family Positive Adaptation Scale. Minimum score=14, maximum score=42. Higher scores correspond to better outcomes.
Therapeutic Alliance | Time 1, 2, 3, 5
  Descriptive (no criterion for success): Working Alliance Inventory-Short Revised (WAI-SR). Minimum score=12, maximum score=60. Higher scores correspond to better outcomes.
Form Research-Clinical Partnership (1) - Clinical-Research Meetings | Time -1 to end of study
  Criterion for success: Meet once monthly throughout the course of the study.
Form Research-Clinical Partnership (2) - Protocol Development - a | Time -1
  Criterion for success: Administrative approval from SKCCMH for study (via approval of ethics approval).
Form Research-Clinical Partnership (3) - Protocol Development - b | Time -1
  Criterion for success: Submission of protocol for registration to clinicaltrials.gov and/or journal publications.
Research-Clinical Communication (1) - Clients Referred to LTP-B | Time -1
  Criterion for success: 95% of clients referred to LTP-B to be asked permission to be contacted by the research team.
Research-Clinical Communication (2) - Clients Transferred to Research Team | Time -1
  Criterion for success: 95% of clients that agree to research are transferred to the research team for contact.
Research-Clinical Communication (3) - Clinical Visits Shared | Time -1 to end of study
  Criterion for success: 95% of participants' scheduled clinical visits to be shared with the research team.
Research-Clinical Communication (4) - Videos Shared | Time 1, 2, 3
  Criterion for success: 95% of participant videos (previously consented) to be successfully shared with the research team.
Clinical Service Flow (1) - Clients Referred | Time -1
  Criterion for success: 3 families to be referred to the LTP-B per month.
Clinical Service Flow (2) - Service Provision | Time -1
  Criterion for success: 2 families to be seen by the LTP-B team per month.
Participant Recruitment (1) - Agree to Research Contact | Time -1
  Criterion for success: 90% of clients referred to LTP-B to agree to be contacted for purposes of research.
Participant Recruitment (2) - Participants Enrolled | Time -1
  Criterion for success: 90% of clients participating in LTP-B to enroll in the research study.
Participant Recruitment (3) Families Enrolled Per Month | Time -1
  Criterion for success: 1.8 families enrolled per month.
Adherence to Intervention | Times 1, 2, 3
  Criterion for success: 90% of participants to complete all three main LTP-B sessions (Family assessment, videofeedback, check in)
Retention: Post-Intervention | Time 3
  Criterion for success: 90% of participants to remain in study until the end of post-intervention assessment.
Retention: Follow-Up | Time 4
  Criterion for success: 80% of participants to remain in study until the end of follow-up assessment.
Retention: Brief Surveys | Time 1, 2, 5
  Criterion for success: 80% of participants to complete all brief surveys.
Acceptability | Time 3, 4
  Criterion for success: 80 % of participants reporting at least "agree" on indicators of attitude, burden, perceived effectiveness, and ethicality on an Implementation Acceptability Scale. Minimum score=7, maximum scores=35. Higher scores correspond to better outcomes.
Descriptive (no criterion for success): Behavioral Coding of Family Interactions (Frascarolo et al., 2018) | Week 1
  Family interactions will be behaviourally coded by trained coders based on the LTP Assessments (initial family assessment), using previously validated approaches (e.g., Frasarolo et al., 2018).

SECONDARY OUTCOMES:
Brief Dyadic Adjustment | Time 0, 1, 2, 3, 4, 5
  Using the Brief Dyadic Adjustment Scale (DAS-4). Minimum score= 0, maximum score=21. Higher scores correspond to better outcomes.
Coparenting Relationship Quality | Time 0, 3, 4
  Using the Brief Coparenting Relationship Scale (Feinberg et al., 2012). Minimum score=0, maximum score=84. Higher scores correspond to better outcomes.
Brief Coparenting Relationship Quality | Time 1, 2, 5
  Using the Subset of Brief Coparenting Relationship Quality Scale (Feinberg et al., 2012). Minimum score=0, maximum score=36. Higher scores correspond to better outcomes.
Parent-Child Positivity | Time 0, 3, 4
  Using the 5-item parent-reported positivity subscale of the Parenting Practices Scale. Minimum score=5, maximum score=25. Higher scores correspond to better outcomes.
Parent-Child Negativity | Time 0, 3, 4
  Using the 5-item parent-reported negativity subscale of the Parenting Practices Scale. Minimum score=5, maximum score=25. Higher scores correspond to worse outcomes.
Sibling Relations | Time 0, 3, 4
  Using Parental Expectations and Perceptions of Children's Sibling Relationship Questionnaire (PEPC-SRQ). Minimum score=8 , maximum score=40. Higher scores correspond to better outcomes.
Whole Family Functioning | Time 0, 3, 4
  Using 6-item Family Assessment Device (FAD). Minimum score=5, maximum score=20. Higher scores correspond to worse outcomes.
Parent Mental Health | Time 0, 3, 4
  Using the Kessler Psychological Distress Scale (K10). Minimum score=10, maximum score=50. Higher scores correspond to worse outcomes.
Brief Parent Mental Health | Time 1, 2, 5
  Using the Kessler Psychological Distress Scale (K6). Minimum score=6, maximum score=30. Higher scores correspond to worse outcomes.
Child Emotional and Behavioural Problems (1) - (Children Ages 18 months to 3 years 11 months) | Time 0, 3, 4
  Scores will be standardized within each age group and used as a single outcome variable.
  The Preschool Pediatric Symptom Checklist (PPSC-17): Minimum score=0, maximum score=36. Higher scores correspond to worse outcomes.
Child Emotional and Behavioural Problems (2) - (Children Ages 4 to 18 years) | Time 0, 3, 4
  Scores will be standardized within each age group and used as a single outcome variable.
  The Pediatric Symptom Checklist (PSC-17). Minimum score=0, maximum score=34. Higher scores correspond to worse outcomes.
Examine Therapy Sessions | Weeks 1, 2, 3
  Examine content and process of all therapy sessions (including therapist and client behaviours) qualitatively for a select number of 'successful' and 'unsuccessful' cases, using a pragmatic case-series analysis (e.g., Liekmeier et al., 2021)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Prime, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided